CLINICAL TRIAL: NCT04488211
Title: Survey of Fertility Specialists' Knowledge of, Experience With, and Attitudes Toward the Use of in Vitro Maturation of Oocytes in Reproductive Medicine
Brief Title: IVM Survey Among Reproductive Medicine Specialists
Status: Completed | Type: Observational
Sponsor: Universitair Ziekenhuis Brussel (Other)
Collaborators: CooperSurgical Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: IVM Survey V2 04062020
Record Dates: First submitted 2020-07-06; First posted 2020-07-27 (Actual); Last update posted 2021-05-04 (Actual); Status verified 2020-06

CONDITIONS: IVM
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Prospective survey respondents: Invitations to participate in the survey will be emailed on three occasions to selected fertility specialists worldwide who are affiliated to a public or private fertility clinic.
  Interventions: Other: Survey

INTERVENTIONS:
Other: Survey — The IVM survey will be structured as a series of open questions and multiple-choice questions.

SUMMARY:
Although IVM as a laboratory technology in reproductive medicine has existed for many decades, there is a lack of well-designed studies comparing the efficiency and the patient satisfaction related to IVM as compared to standard ovarian stimulation for IVF. In view of this, and in order to identify unmet needs of fertility specialists with regard to the application of IVM, the investigator developed the idea of a worldwide web-based survey analysis of fertility specialists' insights and experiences regarding IVM.

DETAILED DESCRIPTION:
The IVM survey will be structured as a series of open questions and multiple-choice questions. In most of the questions, a single answer will be required by participants. A small number of questions will allow multiple answers. The survey will be web-based. Invitations to participate in the survey will be emailed on three occasions to selected fertility specialists worldwide who are affiliated to a public or private fertility clinic. Clinics will be identified based on whether they have worked with IVM previously but stopped, and clinics with appropriate size to offer IVM competence. When no response is obtained from selected fertility specialists, e-mails will be sent to affiliated colleagues working at the same fertility clinic. When analyzing the survey results, care will be taken to analyse the responses per fertility clinic, as responses from different fertility specialists working in the same fertility clinic should be avoided. Results will be analysed using a method that assigns equal weight per clinic and a method that weights clinic responses based on treatment volume (number of IVF cycles).

ELIGIBILITY:
Inclusion Criteria:

* IVF clinics that have worked with IVM previously but stopped
* clinics with appropriate size to offer IVM

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Fertility specialists around the globe who are affiliated to a public or private fertility clinic. Clinics will be identified based on whether they have worked with IVM previously but stopped, and clinics with appropriate size to offer IVM competence.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2020-07-30 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Name of the measurement: Application of in vitro maturation (IVM) of oocytes as a laboratory tool | 1 month
  Measurement tool: questionnaire; unit of measure: % of respondents who use oocyte in vitro maturation in the laboratory;
Name of the measurement: Appreciation of IVM as a laboratory technique | 1 month
  Measurement tool: questionnaire; unit of measure: % of respondents who believe there is a role for IVM in the ART (assisted reproductive technology ) clinic

SECONDARY OUTCOMES:
Name of the measurement: Annual number of egg retrievals for IVM | 1 month
  Measurement tool: questionnaire; unit of measure: number

CONTACTS AND LOCATIONS:
Overall Officials: Michel De Vos, Principal Investigator — Universitair Ziekenhuis Brussel
Locations (1):
- Universitair Ziekenhuis Brussel, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No